CLINICAL TRIAL: NCT03654352
Title: Assessing the Role of Sphingolipids in AcuTE Respiratory Distress Syndrome
Brief Title: The ASTERS Study: Assessing the Role of Sphingolipids in AcuTE Respiratory Distress Syndrome (ARDS)
Acronym: ASTERS
Status: Completed | Type: Observational
Sponsor: Sturgill (Other)
Responsible Party: Sponsor-Investigator, Sturgill, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 44569
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: lung; ceramide; sphingolipid; inflammation; pulmonary; ARDS; ALI
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk for ARDS/ALI: Mechanically ventilated patients with risk factors for the development of ARDS/ALI. These factors are classified into two categories: pulmonary insults, such as pneumonia and extrapulmonary insults such as sepsis.
- Low Risk for ARDS/ALI: Mechanically ventilated patients with low risk factors for the development of ARDS/ALI. These factors include mechanical ventilation for airway protection, pain management, or procedure.

SUMMARY:
Acute lung injury (ALI) and the more severe manifestation, acute respiratory distress syndrome (ARDS) describe syndromes of acute onset, bilateral, inflammatory pulmonary infiltrates and impaired oxygenation. ARDS/ALI are a continuum of disease which results in a life threatening, rapidly progressive illness and occurs in critically ill patients. Recent reports in the Journal of the American Medical Association (JAMA) highlight the significant public health impact ARDS/ALI has on the critically ill population in that despite robust research efforts, these illnesses continue to be under diagnosed, under treated, and continue to have a high mortality rate (≥ 40% of all confirmed diagnoses). The estimates for ARDS/ALI incidence vary due to inconsistencies with proper diagnosis and lack of valid biomarkers of disease; however, it is expected that anywhere from 20-50% of patients on mechanical ventilation will develop this disease. Previous work by our group has shown that sphingolipids play a multifaceted role in lung inflammation. Sphingolipid are a class of bioactive lipids that play a role in cellular processes such as apoptosis, cell migration, and adhesion. Ceramide is one species of sphingolipid the investigators have examined in both man and mouse. Our laboratory has shown that ceramide is up-regulated in pulmonary inflammation in mouse models of pneumonitis and is elevated in the exhaled breath condensate of mechanically ventilated patients at risk for ARDS/ALI. Our work coupled with the work of others highlighting a role for ceramide in chronic obstructive pulmonary disease (COPD), surfactant dysfunction, and infectious disease make ceramide a logical candidate biomarker that warrants further investigation. To our knowledge, there are no studies examining the role of ceramide as a biomarker in ARDS/ALI. Thus, our overarching hypothesis is that ceramide is elevated in the lungs of patients who develop ARDS/ALI. This lipid dysregulation accounts for the pathophysiology seen in this disease and may be a potential pharmacologic target for clinical treatment. Thus the purpose of this exploratory research is to maximize existing specimens to further evaluate ceramide as a biomarker for acute lung injury.

DETAILED DESCRIPTION:
Since it was first described in 1967 by Ashbaugh et al, ARDS/ALI remains a global clinical problem resulting in high morbidity and mortality. These lung syndromes are life threatening, rapidly progressive disease occurring in critically ill patients characterized by hypoxemia, alterations in lung mechanics, and edema. Recent reports in the Journal of the American Medical Association (JAMA) highlight the significant public health impact ARDS/ALI has on the critically ill population in that despite robust research efforts, ARDS continues to be under diagnosed, under treated, and continues to have a high mortality rate (= 40% of all confirmed diagnoses). The estimates for ARDS/ALI incidence vary due to inconsistencies with proper diagnosis and lack of valid biomarkers of disease; however, it is expected that anywhere from 20-50% of patients on long term mechanical ventilation will develop this disease. Despite this robust effort to better improve patient care, clinicians are still lacking biomarkers of disease and a strong understanding of the underlying pathophysiology of ARDS/ALI. Thus, research is warranted in this area. Many research efforts have been aimed at unifying diagnoses of the disease with clinical criteria, thus the ARDS Task force implemented the Berlin definition of disease in 2012 but despite this, recent data from the Lung SAFE trial showed that clinical recognition of disease was only 34.1% on initial presentation, again emphasizing the need for objective measures of disease.

The oxygenation threshold set forth by the Berlin definition are critical for understanding of ARDS/ALI disease severity and progression. Oxygenation is calculated by the PaO2/FiO2 ratio (P/F) which is the the ratio of arterial oxygen partial pressure (PaO2) as determined by arterial blood gas to fractional inspired oxygen setting on the mechanical ventilator (FiO2). This P/F ratio is also important to distinguish both diagnosis of ARDS but disease severity. A normal healthy P/F ratio is between 400-500 whereas ALI is below 300 (aka Mild ARDS by Berlin definition), ARDS is below 200, and severe ARDS is below 100. These are the same clinical parameters used by our medical intensive care unit (MICU). The current treatment modalities for ARDS/ALI are primarily supportive care in the form of lung protective ventilator management, fluid management, prone positioning, and neuromuscular blockage in severe ARDS. Clinical studies have examined potential pharmacologic therapies including the use of albuterol, anti-platelet therapies, statins, aspirin, and steroids - none of which had any significant benefit on clinical outcomes. Our data in mouse models and preliminary data in a small cohort of patients at risk for ARDS/ALI highlight a novel role for ceramide in the pathophysiology of this disease. Our preliminary data indicate that ceramide may not only be a key player in the underlying pathology of ARDS/ALI, but may also serve as a useful biomarker. Additionally, as there is a currently FDA approved drug that targets ceramide formation and actions as the investigators have demonstrated, the work outlined herein has significant translational potential. Thus, this proposal will examine the premise that ceramide is a new critical player in ARDS/ALI and identify ceramide as a biomarker for individualized medicine to optimize diagnosis and improve treatments. Given the large numbers of individuals affected by ARDS/ALI, the outcomes of this research have the potential to change the paradigm of how clinicians and researchers perceive inflammatory airway disease and may then translate into better, targeted approaches for the management for millions worldwide. This pilot study will be conducted as a prospective descriptive, cross-sectional study with a single data collection. This design allows for greater control over the measurements and maximization of data completeness. While a cross-sectional study design does not allow us to examine causality, it does allow us to examine associations among the variables/domains of interest, which align with the aim of the study. This design is appropriate and scientifically rigorous while meeting the budgetary and time constraints of the grant mechanism. The investigators have developed a state of the science, non-invasive technique which can be utilized to assess sphingolipid levels in the breath of mechanically ventilated subjects. Exhaled breath condensate (EBC) is collected using a commercially available device, RTubeVent™ (Respiratory Research Inc., Austin, TX). The RTubeVent™, covered by a frozen aluminum sleeve and fabric cloth sleeve, allows for the cooling of exhaled breath into a condensed liquid form and is a safe, easy, relatively inexpensive, repeatable, non-invasive approach to collect a biological fluid that is hypothesized to be more specific to pulmonary biology changes compared to systemically collected biological fluids such as serum or plasma. The RTubeVENT™ breath condensate collection device is designed for ease of use in the ICU. It can be placed in-line in the expiratory limb of the breathing circuit or at the ventilator exhaust port. This non-invasive device is fully self-contained and disposable. As the subject is ventilated, the RTubeVENT™ gathers breath condensate in a special cartridge designed exclusively for ventilator use. EBC has been identified by the National Institutes of Health as an emerging source for biomarker research thus highlighting another innovative aspect of this proposal. Once patients are enrolled in the study, the investigators will collect EBC from the ventilator for approximately 20 minutes under the guidance of respiratory therapy and take a 5cc blood draw for plasma isolation. Samples will be immediately taken to the laboratory for processing where both EBC and plasma will be aliquoted, and stored at -80°C until analysis. Liquid chromatography electrospray ionization-tandem mass spectrometry (LC-ESI-MS/MS) will be used to detect sphingolipid levels and samples will be batch processed to minimize variability. The investigators predict that patients in the ARDS/ALI group will have significantly elevated ceramide levels as compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

Admission to the medical intensive care unit Mechanically ventilated for less than 48 hours Able to consent in English. -

Exclusion Criteria:

Unable to obtain consent Mechanically ventilated for more than 48 hours Moribund Prisoner or ward of the state Pregnant Less than 18 years old, Metastatic lung cancer.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the medical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Ceramide levels in exhaled breath condensate | We plan to do a single time point data collection. Exhaled breath will be collected for 20 minutes.
  Ceramide is a candidate bio marker we plan to examine to describe patterns of risk factors associated with ARDS/ALI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No